CLINICAL TRIAL: NCT01226342
Title: Transcutaneous Electrical Muscle Stimulation in Acute Exacerbation of Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Transcutaneous Electrical Muscle Stimulation In Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University Clinic of Pulmonary and Allergic Diseases Golnik (Other)
Responsible Party: Principal Investigator, Mitja Lainščak, Professor, The University Clinic of Pulmonary and Allergic Diseases Golnik
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Golnik-COPD-TENS-1
Record Dates: First submitted 2010-10-18; First posted 2010-10-22 (Estimated); Last update posted 2013-04-11 (Estimated); Status verified 2013-04

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Chronic obstructive pulmonary disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TCEMS (Experimental): Patients who will receive transcutaneous electrical muscle stimulation
  Interventions: Device: Transcutaneous electrical muscle stimulation

INTERVENTIONS:
Device: Transcutaneous electrical muscle stimulation — On the first hospitalization day patients received lower extremity TCEMS. We used GymnaUniphy device (GymnaUniphy N.V., 2004, 3740 Bilzen, Belgium) with four surface patch electrodes applied over each lower extremity quadriceps muscle. Patients were in the supine position and were advised to relax during sessions. A prespecified program for lower extremity strength training in sessions of 25 minutes, twice a day (first training in the morning, second in the afternoon, with minimal time difference of 6 hours) was performed six days per week during the hospitalization.

SUMMARY:
Transcutaneous electrical muscle stimulation (TCEMS) is well established intervention for rehabilitation of clinically stable patients with chronic obstructive pulmonary disease.

The investigators have conceived this study to test whether TCEMS is feasible and tolerated by patients experiencing severe physical and psychical challenge of acutely exacerbated COPD.

ELIGIBILITY:
Inclusion Criteria:

* chronic obstructive pulmonary disease GOLD stage III or IV
* acute exacerbation of the disease

Exclusion Criteria:

* contraindications for transcutaneous electrical muscle stimulation

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2009-01; Primary Completion 2009-06 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Scores on the feasibility scale | 10 days (avarage time from admission to discharge)
  Patients will be followed from admission until discharge

SECONDARY OUTCOMES:
Scores on the patient satisfaction scale | 10 days (avarage time from admission to discharge)
  Patients will be followed from admission until discharge
Number of patients with adverse events as a measure of Safety and tolerability | 10 days (avarage time from admission to discharge)
  Patients will be followed from admission until discharge
Health related quality of life on the St. George respiratory questionnaire | 10 days (avarage time from admission to discharge)
  Patients will be followed from admission until discharge
Dyspnea on the MRC dyspnea scale | 10 days (avarage time from admission to discharge)
  Patients will be followed from admission until discharge
Patient symptom scores on the Functional assessment of chronic illness therapy questionaire | 10 days (avarage time from admission to discharge)
  Patients will be followed from admission until discharge

CONTACTS AND LOCATIONS:
Overall Officials: Mitja Lainscak, MD, PhD, Principal Investigator — University Clinic Golnik; Mitja Kosnik, MD, PhD, Study Chair — contraindications for TCEMS
Locations (1):
- University Clinic Golnik, Golnik, Slovenia

REFERENCES:
- [Result] Meglic U, Sorli J, Kosnik M, Lainscak M. Feasibility of transcutaneous electrical muscle stimulation in acute exacerbation of COPD. Wien Klin Wochenschr. 2011 Jun;123(11-12):384-7. doi: 10.1007/s00508-011-1587-2. Epub 2011 May 25. PMID 21607562